CLINICAL TRIAL: NCT02923128
Title: Whether Dexmedetomidine Can Improve the Prognosis of Elderly Patients With Postoperative Cognitive Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xie Kangjie, MD, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-01-13
Record Dates: First submitted 2016-09-11; First posted 2016-10-04 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium | interventions — Dexmedetomidine; Sufentanil; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine+routine PCIA (Active Comparator): PCIA pump was provided after surgery, which consisted of 3 ug/kg sufentanil and 3 ug/kg dexmedetomidine, total amount 150ml, 2 mL bolus dose with a lock-out of 10 minutes and background infu-sion rate 2 mL/h.
  Interventions: Drug: Dexmedetomidine; Drug: Sufentanyl; Drug: Saline
- Routine PCIA (Sham Comparator): 3 ug/kg sufentanil without dexmedetomidine, total amount 150ml, 2 mL bolus dose with a lock-out of 10 minutes and background infu-sion rate 2 mL/h.
  Interventions: Drug: Sufentanyl; Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 3 ug/kg is diluted to 150ml with 0.9% saline,continuous micro-pump infusion for 72 hours with 2ml/h speed.
  Other Names: Dexmedetomidine Hydrochloride Injection
  Arms: Dexmedetomidine+routine PCIA
Drug: Sufentanyl — Sufentanyl 3 ug/kg is diluted to 150ml with 0.9% saline,continuous micro-pump infusion for 72 hours with 2ml/h speed.
  Other Names: Sufentanil Citrate Injection
Drug: Saline — Saline is used to dilute other drugs
  Other Names: normal saline,physiological saline,NS

SUMMARY:
The purpose of this study is to determine whether postoperative analgesia pump continuous infusion of dexmedetomidine are effective in the prevention of Postoperative delirium and Postoperative cognitive dysfunction.

DETAILED DESCRIPTION:
1. collection of cases: This trail is approved by Hospital Ethics Committee, and patients who participated in the study signed the informed consent. The subject will select 300 elder patients (age ≥60 years) routine tumor surgery, American Society of Anesthesiologists classificationⅠ-Ⅲ. Preoperative liver and kidney function, blood electrolytes were in the normal range.
2. Case group: Selected cases divided into the right dexmedetomidine group and control group by computer randomly, 150 patients in each group. Dexmedetomidine group (A group) analgesia pump formula is: 3 ug/kg sufentanil and 3 ug/kg dexmedetomi-dine, with 0.9% saline diluted to 150ml. Control group (group C) postoperative analgesia formula is: 3 ug/kg sufentanil, with 0.9% saline diluted to 150ml. Two group with the same anesthesia program.
3. Our primary outcome was the 7-day incidence of postoperative delirium assessed by CAM-ICU twice daily (8 a.m. and 8 p.m.) and supplemented with a review of medical and nursing records. The assessment was carried out by investigators who had been trained prior to the trial and were unaware of the group assignment.All investigators and patients were unknown of experiments and results. The four clinical criteria for CAM-ICU are as follows: (1) acute onset with fluctuating course of disease; (2) inattention; (3) altered level of consciousness; (4) disorganized thinking. Delirium can be diagnosed by the appearance of both features 1 and 2, with at least one of features 3 or 4. RASS was used to measure sedation or agita-tion prior to testing delirium. If the patient was deeply sedated or unable to fall asleep (RASS - 4 or - 5), delirium assessment was halted; if RASS score was of - 3 or above, delirium was evaluated by CAM-ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age ≥60 years
* Underwent elective non-cardiac surgery under general anesthesia

Exclusion Criteria:

* Patients with severe bradycardia (heart rate<55bpm)
* Severe arrhythmia or cardiac dysfunction (ejection fraction<35%)
* Mini-Mental Scale Test (MMSE) Exclusion criteria: illiteracy <18, primary school <21, junior school and above <25
* Preoperative clear systems and spiritual history of neurological disease or long-term use of sedatives or antidepressants
* History of alcohol abuse or a history of drug dependence
* Have brain surgery or trauma
* Severe vision or hearing impairment
* Cannot with the completion of tests of cognitive function
* Refused to participate in the study

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 7 days after surgery
  The four clinical criteria for CAM-ICU are as follows: (1) acute onset with fluctuating course of disease; (2) inattention; (3) altered level of consciousness; (4) disorganized thinking. Delirium can be diagnosed by the appearance of both features 1 and 2, with at least one of features 3 or 4.

SECONDARY OUTCOMES:
NRS for pain | 3 days after surgery
  Pain was assessed by NRS (Numeric Rating Scale) : assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable".
Adverse events | 3 days after surgery
  including hypotension, hypertension, bradycardia, tachycardia, hypoxemia, and in-terventions (adjustment or stop study drug infusion or intravenous administration).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No